CLINICAL TRIAL: NCT01467128
Title: Title of Study: Adverse Drug Event (ADE) Incidence in Older Patients Following Hospital Admission and Pharmacist Review to Older Persons' Prescriptions and Its' Effect on ADE Reduction in Hospital: a Randomised Controlled Trial
Brief Title: Adverse Drug Event Prevention Using Structured Pharmacist Review
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Denis O'Mahony, Senior Lecturer, Dept. of Medicine, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HRA_HSR/2010/14(a)
Record Dates: First submitted 2011-09-02; First posted 2011-11-08 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Adverse Drug Reactions
Keywords: Elderly; Hospital; Adverse Drug; Pharmacist; Prevention
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured expert pharmacist review (Active Comparator)
  Interventions: Other: Structured expert pharmacist review
- Normal pharmaceutical care in hospital (No Intervention)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Structured expert pharmacist review — The researcher will apply the pharmacist intervention to the cases randomised to this arm of the study. This consists of an expert pharmacist review of the patients prescribed medications at the time of recruitment into the study. Recommendations following the intervention will be communicated both verbally and in writing to the medical team with primary responsibility for the patient. Recommendations arising from the intervention will be printed out and inserted into the patients' notes, in addition to the relevant registrar being informed in person or via the telephone.
  Other Names: expert pharmacist review
  Arms: Structured expert pharmacist review
Other: No Intervention — Normal hospital pharmaceutical care
  Arms: Normal pharmaceutical care in hospital

SUMMARY:
The next four decades will see a marked expansion of the elderly population in Ireland, in particular people aged over 80 yrs. Persons aged over 80 are the highest consumers of prescription medicines in Ireland and have the highest prevalence rates of major polypharmacy. Polypharmacy is intimately linked with serious adverse drug events (ADEs) and consequent major morbidity and mortality. Epidemiological data from the Unites States indicate that ADEs is the fifth most common cause of death nationally. Experts suggest that effective evidence based interventions can be applied to this major public health problem.

A recently described approach to hospitalised older patients' medication optimisation is that of Spinewine and colleagues at Louvain University, Belgium. In this model, a pharmacist with expertise in geriatric pharmacotherapy routinely reviews the prescriptions of older patients from admission to discharge. The pharmacist provides a detailed pharmaceutical care plan for older patients and their carers where appropriate as well as feedback information to prescribers in the event of detecting instances of probable medication inappropriateness. Whenever an opportunity for medication optimisation is identified, the pharmacist discusses the opportunity with the prescriber who can accept or reject the intervention. At discharge from hospital, the pharmacist also provides written and verbal information on treatment changes to the patient / caregiver and GP. The intervention therefore represents a comprehensive pharmaceutical care approach that is based upon careful review and subsequent consensus on individualised pharmacotherapy. In an RCT comparison of this approach with standard care, older patients in the intervention arm of the study had significant improvements in medication appropriateness (medication appropriateness index (MAI), Beers' criteria, and Assessing Care of Vulnerable Elders (ACOVE) criteria.). Expert pharmacist review of older peoples' medication in hospital is a proven intervention in term of reducing inappropriateness of medication.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 65 years and over presenting to CUH Accident and Emergency Departments with acute illness for admission under a medical team will be eligible for the study.

Exclusion Criteria:

1. Age less than 65 years.
2. Patient to be admitted under the care of a Geriatrician Psychiatrist of Old Age or Clinical Pharmacologist, or having been admitted under these services or attended their outpatient clinics in the previous 12 months. (These doctor groups are likely to minimise inappropriate medications in this population).
3. Terminally ill patient attended by palliative care team.
4. Critically ill patient e.g. admitted to Intensive Care Unit.
5. Patients who do not wish to participate in the study.
6. Patients whose hospital physician does not wish to participate in the study ver, its efficacy in terms of ADE prevention is not yet demonstrated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 720 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with definite and possible adverse drug events during their hospital admission | From point of randomization to Day 14

SECONDARY OUTCOMES:
Drug ingredient cost at hospital discharge | Up to Day 14
Medication Appropriateness Index score | measured at Day 14 and again at three months post hospital discharge.
Composite health resource utilization including hospital admissions and primary care consultations | Measured at 3 months post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: David O'Sullivan, MPharm, Study Director — University College Cork, Ireland
Locations (1):
- Cork University Hospital, Cork, Munster, Ireland

REFERENCES:
- [Background] Spinewine A, Dhillon S, Mallet L, Tulkens PM, Wilmotte L, Swine C. Implementation of ward-based clinical pharmacy services in Belgium--description of the impact on a geriatric unit. Ann Pharmacother. 2006 Apr;40(4):720-8. doi: 10.1345/aph.1G515. Epub 2006 Mar 28. PMID 16569792
- [Background] Spinewine A, Swine C, Dhillon S, Lambert P, Nachega JB, Wilmotte L, Tulkens PM. Effect of a collaborative approach on the quality of prescribing for geriatric inpatients: a randomized, controlled trial. J Am Geriatr Soc. 2007 May;55(5):658-65. doi: 10.1111/j.1532-5415.2007.01132.x. PMID 17493184
- [Background] Hamilton H, Gallagher P, Ryan C, Byrne S, O'Mahony D. Potentially inappropriate medications defined by STOPP criteria and the risk of adverse drug events in older hospitalized patients. Arch Intern Med. 2011 Jun 13;171(11):1013-9. doi: 10.1001/archinternmed.2011.215. PMID 21670370
- See also: Health Research Board (Ireland) website — http://hrb.ie